CLINICAL TRIAL: NCT03704636
Title: Desaturation Validation of INVSENSOR00028
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19457
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00028 sensor.
  Interventions: Device: INVSENSOR00028

INTERVENTIONS:
Device: INVSENSOR00028 — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to measure the trending accuracy of a noninvasive regional oximetry measurement of somatic oxygen saturation. Two large sensors (adult sensors) will be placed on the subject's forehead. Two investigational sensors (INVSENSOR00028) will be placed on the forearm of the volunteer. The values obtained by the INVSENSOR00028 will be compared to the reference value calculated from the arterial and venous blood measurements. Data will be collected from healthy adult subjects while undergoing a desaturation procedure wherein the concentration of oxygen inhaled is slowly reduced until the subject's arterial oxygen saturation is approximately 70%, while blood samples are drawn at prespecified reference points. The subject will then be returned to inhaling room air.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* CO value ≤ 2.0% FCOHb
* Subject has a physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Systolic Blood Pressure ≤ 140 mmHg and Diastolic Blood Pressure ≤ 90 mmHg.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant.
* Subject smokes (smoking includes e-cigarette use).
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after a blood draw.
* Subject has open wounds, inflamed tattoos or piercings, visible healing wounds.
* Subject experiences frequent or severe headaches and/or migraine headaches.
* Subject has known drug or alcohol abuse and/or use of recreational drugs.
* Subject has experienced a concussion or head injury with loss of consciousness within the last year.
* Subject has any chronic bleeding disorders (i.e. hemophilia).
* Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
* Subject has any cancer or history of cancer (not including skin cancer).
* Subject has a chronic neurological disease (i.e. multiple sclerosis, Huntington's Disease).
* Subject has any cardiac dysrhythmia(s) (i.e. atrial fibrillation) and has not received clearance by their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subject's level of consciousness.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator).
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject who has taken anticoagulant medication within the last 30 days.
* Subject has taken opioid pain medication within 24 hours of start of study.
* Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, plastic surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has donated blood within the past 30 days.
* Subject has symptoms of congestion, head colds, flu or other illnesses.
* Subject experiences claustrophobia or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent diabetes or uncontrolled hypertension.
* Subject has given vaginal delivery, had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
* Subject intends to participate in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours of the study.
* Discretion of investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 46 enrolled participants, 23 met inclusion criteria and proceeded to the study. The remainder of the enrolled participants include screen failures and subjects that did not proceed due to time constraints.
Period: Overall Study
Arm/Group | Test Subject
Started | 23
Completed | 20
Not Completed | 3
Not completed — Inadequate Venous Flow | 3

BASELINE CHARACTERISTICS:
Arm/Group | Test Subject
Number analyzed (Participants) | 20
Age, Customized [Count of Participants; unit: Participants]
  < 18 years old | 0
  18 to 50 years old | 20
  > 50 years old | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 2
  Caucasian | 8
  Black or African American | 6
  Hispanic | 4

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation (rSO2) Accuracy of Sensor
Description: The Trending accuracy of the INVSENSOR00028 will be evaluated relative to the reference value calculated from the arterial and venous blood measurements.
Time Frame: 1-5 hours
Population: There is no apparent trend in either the Brachial or Flexor RSO2 data with respect to the control. Since there is no measurable trend, a numerical value for Trending Accuracy (as defined in the protocol) cannot be accurately determined.
Arm/Group | Test Subject
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 to 5 hours
Arm/Group | Test Subject
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Subject (N=20)
Hematoma (Injury, poisoning and procedural complications) | 1
Sensitivity at arterial line site (Injury, poisoning and procedural complications) | 1
Lightheadedness (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03704636/Prot_SAP_000.pdf